CLINICAL TRIAL: NCT03415191
Title: Is The Pre-Emptive Administration Of Ketamine A Significant Adjunction To Intravenous Morphine Analgesia For Controlling Post-Operative Pain? A Randomized, Double Blind, Placebo Controlled Clinical Trial.
Brief Title: The Pre-Emptive Administration Of Ketamine for Controlling Post-thoracotomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Alfonso Fiorelli, Assistant Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 513/12
Record Dates: First submitted 2018-01-15; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Post Thoracotomy Pain
Keywords: ketamine, post-thoracotomy pain, analgesia
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This was a single center, double-blind, placebo controlled, parallel-group, prospective study. Patients were randomly assigned to Ketamine or Placebo group in 1:1 ratio and no changes to methods after trial commencement as type of randomization or eligibility criteria were attended.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Experimental): Five minutes before thoracotomy incision, Ketamine Group received a bolus dose of ketamine 1 mg/kg intravenously
  Interventions: Drug: Ketamine
- Placebo Group (Placebo Comparator): Five minutes before thoracotomy incision, Placebo Group received a bolus dose of normal saline 1 mg/kg intravenously
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ketamine — A bolus dose of ketamine 1 mg/kg intravenously five minutes before surgical incision
  Arms: Ketamine Group
Drug: Normal Saline — A bolus dose of normal saline 1 mg/kg intravenously five minutes before surgical incision
  Arms: Placebo Group

SUMMARY:
The goal of this paper is to evaluate whether the pre-emptive administration of Ketamine would potentiate the effect of intravenous morphine analgesia in management of post thoracotomy pain. This was a single center, double-blind, placebo controlled, parallel-group, prospective study. Patients were randomly assigned to receive 1 mg/kg ketamine (Ketamine Group) or an equivalent dose of normal saline (Placebo Group) before thoracotomy in 1:1 ratio. All patients received postoperatively intravenous morphine administration as additional analgesic regimen Primary end-point was pain relief measured with Visual Analogue Scale at rest. The secondary end-points were the reduction of inflammatory response expressed by plasma c-reactive protein levels, the morphine consumption, and the rate of side effects. The measurements were carried out 6; 12; 24; 36; and 48 post operative hours.

DETAILED DESCRIPTION:
Thoracotomy is one of the most painful surgical incision. Inadequate control of pain can have several detrimental effects, including increased postoperative morbidity and delayed recovery as well as occurrence of post thoracotomy syndrome. Therefore, choosing an effectiveness analgesic regimen for thoracic surgery is critical. Many strategies including intercostal nerve block, intra pleural analgesia, lumbar or thoracic epidural, paravertebral block, intra venous narcotics, intrathecal or epidural narcotics or trans-cutaneous nerve stimulation have been used with varied success. However, the ideal strategy remains an open issue. Different factors including trauma of chest wall, thoracic viscera, diaphragm, and intercostal nerves concur to thoracotomy pain development. Thus, due to multifactorial genesis of pain following thoracotomy a multimodal analgesic approach rather than a single method seems to be more effective because it blocks noxious input at different targets and levels of pain pathways.

Ketamine is an antagonist of N-methyl-D-aspartate (NMDA) receptor that not only abolishes peripheral afferent noxious stimulation, but it may also prevent central sensitization of nociceptors as shown in animal studies. In thoracic surgery, there are contradictory results on the efficacy of ketamine for controlling pain due to different dose, type of surgery/patient, and postoperative analgesic regimen used in the various studies. Mathew et al. in a recent review concluded that adding low-dose ketamine to intravenous morphine analgesia following thoracotomy was safe and could provide a significant better pain relief and reduction of morphine consumption compared to placebo. D'Alonzo et al. found that the administration of a single dose of ketamine prior to chest incision failed to significantly reduce the pain scores and inflammation in the first 24 post-operative hours. Similarly, Yazigi et al. reported that pre-emptive intravenous low-dose ketamine followed by continuous administration during surgery did not decrease acute pain scores and supplemental morphine consumption. Other studies reported that the epidural infusion of Ketamine before thoracotomy or during thoracic surgery provides better postoperative analgesia compared to placebo group or epidural ropivacaine group In the present study, the investigators supposed that the pre-emptive administration of Ketamine would potentiate the effect of intravenous opioid analgesia with reduction of pain scores, inflammatory response and morphine consumption without increasing morbidity in patients undergoing thoracotomy.

This was a single center, double-blind, placebo controlled, parallel-group, prospective study. Patients were randomly assigned to receive 1 mg/kg ketamine (Ketamine Group) or an equivalent dose of normal saline (Placebo Group) before thoracotomy in 1:1 ratio. All patients received postoperatively intravenous morphine administration as additional analgesic regimen Primary end-point was pain relief measured with Visual Analogue Scale at rest. The secondary end-points were the reduction of inflammatory response expressed by plasma c-reactive protein levels, the morphine consumption, and the rate of side effects. The measurements were carried out 6; 12; 24; 36; and 48 post operative hours.

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 years old,
* planned for an elective partial pneumonectomy (partial or total lobectomy involving one or more lobes, except total pneumonectomy)
* standard lateral thoracotomy for management of non small cell lung cancer (NSCLC)

Exclusion Criteria:

* allergy to Ketamine
* ASA score more than 3
* previous thoracic surgical procedures or lung resection
* mental disease
* participation to other studies
* lack of written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2014-12-21 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Pain Scores on the Visual Analog Scale at 48 hours | 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours after suregry
  The primary end-point was to evaluate whether ketamine was able to reduce the postoperative pain at the first 48 post-operative hours, compared to placebo. The pain levels were scored using a Visual Analogue scale (VAS) ranging from 0=absence of pain to 10= maximal level of pain.

SECONDARY OUTCOMES:
Change From Baseline in c-Reactive Protein (CRP) serum levels at 48 hours | 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours following surgery.
  The inflammatory response was represented by the measurements of c-Reactive Protein (CRP) serum levels in both arms
Change From Baseline in morphine consumption at 48 hours | 6 hours, 12 hours, 24 hours, 36 hours, and 48 hours of postoperative course.
  Cumulative dose of morphine consumption (in mg) was registered in post-operative course
Indicence of clinical adverse effect in the entire post operative course | entire post-operative course
  blurred vision, hallucination, nightmares, vertigo, or nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Fiorelli, MD, PhD, Principal Investigator — University of Campania Luigi Vanvitelli
Locations (1):
- Alfonso Fiorelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romero A, Garcia JE, Joshi GP. The state of the art in preventing postthoracotomy pain. Semin Thorac Cardiovasc Surg. 2013 Summer;25(2):116-24. doi: 10.1053/j.semtcvs.2013.04.002. PMID 24216528
- [Background] Fiorelli A, Vicidomini G, Laperuta P, Busiello L, Perrone A, Napolitano F, Messina G, Santini M. Pre-emptive local analgesia in video-assisted thoracic surgery sympathectomy. Eur J Cardiothorac Surg. 2010 Mar;37(3):588-93. doi: 10.1016/j.ejcts.2009.07.040. Epub 2009 Sep 12. PMID 19748277
- [Background] Burton AW, Lee DH, Saab C, Chung JM. Preemptive intrathecal ketamine injection produces a long-lasting decrease in neuropathic pain behaviors in a rat model. Reg Anesth Pain Med. 1999 May-Jun;24(3):208-13. doi: 10.1016/s1098-7339(99)90129-3. PMID 10338169
- [Background] Lee IO, Lee IH. Systemic, but not intrathecal, ketamine produces preemptive analgesia in the rat formalin model. Acta Anaesthesiol Sin. 2001 Sep;39(3):123-7. PMID 11688102
- [Background] Mathews TJ, Churchhouse AM, Housden T, Dunning J. Does adding ketamine to morphine patient-controlled analgesia safely improve post-thoracotomy pain? Interact Cardiovasc Thorac Surg. 2012 Feb;14(2):194-9. doi: 10.1093/icvts/ivr081. Epub 2011 Nov 28. PMID 22159259
- [Background] Joseph C, Gaillat F, Duponq R, Lieven R, Baumstarck K, Thomas P, Penot-Ragon C, Kerbaul F. Is there any benefit to adding intravenous ketamine to patient-controlled epidural analgesia after thoracic surgery? A randomized double-blind study. Eur J Cardiothorac Surg. 2012 Oct;42(4):e58-65. doi: 10.1093/ejcts/ezs398. Epub 2012 Jul 12. PMID 22790008
- [Background] Tena B, Gomar C, Rios J. Perioperative epidural or intravenous ketamine does not improve the effectiveness of thoracic epidural analgesia for acute and chronic pain after thoracotomy. Clin J Pain. 2014 Jun;30(6):490-500. doi: 10.1097/AJP.0000000000000005. PMID 24281290
- [Background] D'Alonzo RC, Bennett-Guerrero E, Podgoreanu M, D'Amico TA, Harpole DH, Shaw AD. A randomized, double blind, placebo controlled clinical trial of the preoperative use of ketamine for reducing inflammation and pain after thoracic surgery. J Anesth. 2011 Oct;25(5):672-8. doi: 10.1007/s00540-011-1206-4. Epub 2011 Aug 2. PMID 21809148
- [Background] Yazigi A, Abou-Zeid H, Srouji T, Madi-Jebara S, Haddad F, Jabbour K. The effect of low-dose intravenous ketamine on continuous intercostal analgesia following thoracotomy. Ann Card Anaesth. 2012 Jan-Mar;15(1):32-8. doi: 10.4103/0971-9784.91479. PMID 22234019
- [Background] Suzuki M, Haraguti S, Sugimoto K, Kikutani T, Shimada Y, Sakamoto A. Low-dose intravenous ketamine potentiates epidural analgesia after thoracotomy. Anesthesiology. 2006 Jul;105(1):111-9. doi: 10.1097/00000542-200607000-00020. PMID 16810002
- [Background] Feltracco P, Barbieri S, Rizzi S, Ori C, Groppa F, De Rosa G, Frigo AC, Padrini R. Brief report: perioperative analgesic efficacy and plasma concentrations of S+ -ketamine in continuous epidural infusion during thoracic surgery. Anesth Analg. 2013 Jun;116(6):1371-5. doi: 10.1213/ANE.0b013e31828cbaf0. Epub 2013 Apr 4. PMID 23558843